CLINICAL TRIAL: NCT05727215
Title: Immunogenicity and Safety of IndoVac® as a Heterologous Booster Dose Against COVID-19 in Children 12-17 Years of Age
Brief Title: Heterologous Booster Study of COVID-19 Protein Subunit Recombinant Vaccine in Children 12-17 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CoV2-Booster-Children-0222
Record Dates: First submitted 2023-02-13; First posted 2023-02-14 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine; healthy population; Booster; Heterologous; Children
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary dose of inactivated (Sinovac®) vaccine (Experimental): Subject who had received a complete primary dose of inactivated (Sinovac®) vaccine
  Interventions: Biological: SARS-CoV-2 subunit protein recombinant vaccine

INTERVENTIONS:
Biological: SARS-CoV-2 subunit protein recombinant vaccine — SARS-CoV-2 RBD subunit recombinant protein, manufactured by PT. Bio Farma

SUMMARY:
The goal of this clinical trial is to evaluate immune response and safety of SARS-CoV-2 subunit protein recombinant vaccine (IndoVac) as a heterologous booster dose in healthy children 12-17 years of age.

Participants who had received complete primary doses of inactivated (Sinovac®) COVID-19 Vaccine will be given IndoVac as a booster dose.

DETAILED DESCRIPTION:
This trial is open label prospective intervention study. In this study 150 subjects who had received complete primary doses of inactivated (Sinovac®) COVID-19 Vaccine and willing to participate in the booster study by signing the consent form, will be involved in this trial.

Subject will receive one booster dose of SARS-CoV-2 subunit protein recombinant vaccine (IndoVac).

ELIGIBILITY:
Inclusion Criteria:

1. Clinically healthy children 12-17 years of age.
2. Subjects who have previously received complete primary series of inactivated (Sinovac®) COVID-19 vaccine with the last dose administered a minimum of 6 months prior to inclusion but not longer than 12 months prior to inclusion.
3. Parent/legal guardian and subject has been informed properly regarding the study, and signed the informed consent form (parent/legal guardian) and assent form (subject).
4. Parent and/or legal guardian will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

1. Subject concomitantly enrolled or scheduled to be enrolled in another trial.
2. Subject who has received booster dose of COVID-19 vaccine.
3. Subject who has history of COVID-19 in the last 3 months (based on anamnesis or other examinations).
4. Evolving mild, moderate or severe illness, especially infectious disease or fever (body temperature ≥37.5℃, measured with infrared thermometer/thermal gun).
5. History of uncontrolled asthma, history of allergy to vaccines or vaccine ingredients, and severe adverse reactions to vaccines, such as urticaria, dyspnea, and angioneurotic edema.
6. History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
7. Patients with serious chronic diseases (serious cardiovascular diseases, uncontrolled hypertension and diabetes, liver and kidney diseases, malignant tumors, etc) which according to the investigator might interfere with the assessment of the trial objectives.
8. Subjects who have any history of confirmed or suspected immunosuppressive or immunodeficient state, or received in the previous 4 weeks a treatment likely to alter the immune response (intravenous immunoglobulins, blood-derived products or long-term corticosteroid therapy (> 2 weeks)).
9. Subjects who have history of uncontrolled epilepsy or other progressive neurological disorders, such as Guillain-Barre Syndrome.
10. Subjects receive any vaccination (other than COVID-19 vaccine) within 1 month before and after IP immunization.
11. Female who are pregnant or planning to become pregnant during the study period (judged by self-report of subjects and urine pregnancy test results).
12. Subjects plan to move from the study area before the end of study period.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of the candidate vaccine | 14 days after booster vaccination
  Geometric Mean Titer (GMT) and GMFR of neutralizing antibody to the SARS-CoV-2

SECONDARY OUTCOMES:
Seropositive rate of the candidate vaccine | baseline, 14 days, 3 months, 6 months, and 12 months after booster vaccination
  Seropositive rate of neutralizing antibody
Seroconversion rate of the candidate vaccine | baseline and 14 days after booster vaccination
  Seroconversion rate of neutralizing antibody
Seropositive rate and GMT of candidate vaccine | baseline, 14 days, 3 months, 6 months, and 12 months after booster vaccination
  Seropositive rate and GMT of IgG antibody (RBD)
Seroconversion rate of candidate vaccine | baseline and 14 days after booster vaccination
  Seroconversion rate of IgG antibody (RBD)
Safety of the candidate vaccine | 30 minutes, 7 days, 28 days, and until 12 months after booster vaccination
  Percentage of subjects with solicited and unsolicited Adverse Events (AE)
Serious Adverse Event (SAE) of the vaccine | until 12 months after booster vaccination
  Percentage of subjects with at least 1 SAE

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Fadlyana, MD, Principal Investigator — Universitas Padjadjaran
Locations (1):
- Faculty of Medicine Universitas Padjadjaran, Bandung, West Java, Indonesia